CLINICAL TRIAL: NCT03731273
Title: Compensation for Smaller Portion Sizes and Portion Size Normality: Two Laboratory
Brief Title: Compensation for Smaller Portion Sizes and Portion Size Normality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Eric Robinson, Senior Lecturer, University of Liverpool
Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Portion size normality
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Portion Size
MeSH Terms: interventions — Portion Size

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: portion size — Smaller than normal portion size - the intervention is the meal size perceived as 'smaller than normal' that participants are provided with during a lunchtime session in the laboratory.
  'Small-normal' portion size - the intervention is the meal size perceived as 'small normal' that participants are provided with during a lunchtime session in the laboratory.
  'Large normal' portion size - the intervention is the meal size perceived as 'large normal' that participants are provided with during a lunchtime session in the laboratory.

SUMMARY:
Reducing food portion size is a potential strategy to reduce energy intake. However it is unclear at what point consumers compensate for reductions in portion size by increasing energy intake from other items. The investigators tested the hypothesis that reductions to food portion size will only result in significant compensatory eating when the reduced portion size is no longer visually perceived as 'normal'. In two within-subjects experiments, participants (Study 1: N = 45, M BMI = 26.9; Study 2: N = 37, M BMI = 26.9; 51% female) were served different sized portions of a lunchtime meal on three occasions: a 'large-normal', a 'small-normal', and a 'smaller than normal' portion. Both the reduction from 'large-normal' to 'small-normal' and from 'small-normal' to 'smaller than normal' portions represented the same change in food volume and energy content (84g, 77kcal Study 1; 98g, 117kcal Study 2). Participants were able to serve themselves additional helpings of the same food (Study 1), or dessert items (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* general liking and willingness to consume the test foods in each study

Exclusion Criteria:

* food allergies, intolerances or specific dietary requirements (including being vegetarian or vegan)
* a history of eating disorders;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Meal energy intake | Immediate
  Energy intake from the served portion
'Compensatory' (additional) energy intake | Immediate
  Energy intake from additional food provided for consumption after the portion-manipulated meal

CONTACTS AND LOCATIONS:
Locations (1):
- Ashleigh Haynes, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD is available on the Open Science Framework https://osf.io/txf9u/